CLINICAL TRIAL: NCT01992016
Title: A Pilot Study to Enhance F18 FDG-PET Imaging of Prostate Cancers With the Metabolic Inhibitor Ranolazine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-1908.cc; NCI-2013-02000 (Other: National Cancer Institute)
Record Dates: First submitted 2013-11-12; First posted 2013-11-25 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Adenocarcinoma of the Prostate; Bone Metastases; Soft Tissue Metastases; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
Keywords: Prostate cancer; F18 FDG-PET; Imaging; Ranolazine; Bone metastases; Soft tissue metastases
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (localized prostate cancer) (Experimental): Patients receive ranolazine PO BID for 1 day. Patients undergo FDG-PET/CT scan at baseline and after ranolazine treatment. Patients may then undergo robotic or open radical prostatectomy.
  Interventions: Drug: Ranolazine
- Arm II (metastatic prostate cancer) (Experimental): Patients receive ranolazine PO BID for 1 day. Patients undergo FDG-PET/CT scan at baseline and after ranolazine treatment.
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — 1000mg given orally twice daily for 1 day (2 doses).
  Other Names: Ranexa

SUMMARY:
This pilot clinical trial studies fludeoxyglucose F18 (FDG)-positron emission tomography (PET) in imaging patients with prostate cancer treated with ranolazine. Diagnostic procedures, such as FDG-PET, may help find prostate cancer and find out how far the disease has spread. Giving ranolazine may enhance FDG-PET imaging by increasing the amount of glucose available for uptake by the scan.

DETAILED DESCRIPTION:
PET scans have traditionally not been very good at detecting prostate cancers. This is because prostate cancer cells do not take up glucose well so the signals are very weak. The ability of PET imaging to detect cancers requires that the cancer cells take up glucose into the cells. Different methods are being tested to see if we can improve the detection of prostate cancers using PET scans.

Ranolazine is a drug that is already approved by the FDA for treatment of chronic chest pain in people with heart disease. Ranolazine has been studied in the laboratories at the University of Colorado Denver, Anschutz Medical Campus. Ranolazine has been added to prostate cancer cells and grown in petri dishes and in animals in the laboratory. It has been shown to increase the glucose uptake of prostate cancer cells. The goal of this study is to see if patients taking ranolazine will have better PET imaging of their prostate cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained.
2. Adults over 18 years of age.
3. Histological or cytologically confirmed prostate adenocarcinoma.
4. Arm 1 patients must have treatment-naïve, Gleason ≥ 7 prostate cancer based on transrectal ultrasound (TRUS) biopsy, have localized disease, and have decided to undergo radical prostatectomy (open or robotic) as definitive treatment for their prostate cancer.
5. Arm 2 patients must have lymph node, soft tissue, bone, or visceral metastatic disease measuring ≥ 1 cm (lytic component if bone), documented by either CT or MRI imaging within 6 weeks of signing consent. Arm 2 patients may have hormone-sensitive or castrate-resistant disease and may be receiving treatment with hormonal therapies.
6. For Arm 1 patients, the time from the TRUS prostate biopsy to the planned first study PET scan must be ≥ 1 month. For patients who have undergone prior prostate mapping biopsy, the time from the mapping biopsy to the planned first study PET scan must be ≥ 2 months.
7. For Arm 1 patients, participation in this study, in the opinion of the treating physicians, will not introduce delays in surgery that would adversely affect the patient.
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
9. Fasting blood glucose ≤ 120 mg/dL.
10. Adequate renal function (Creatinine ≤ 1.5 X ULN)
11. Adequate hepatic function (bilirubin < 1.5 X upper limit of normal (ULN), alanine aminotransferase (ALT) < 1.5 X ULN, aspartate aminotransferase (AST) < 1.5 X ULN, and albumin ≥ 3 g/dL. For patients with known bone metastases, alkaline phosphatase < 5 X ULN is acceptable.
12. Must be able to take oral medication without crushing, dissolving or chewing tablets.
13. Written authorization for use and release of health and research study information has been obtained.
14. Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection during the study and for 1 week after the last dose of ranolazine.

Exclusion Criteria:

1. Have small cell carcinoma or neuroendocrine component >50%.
2. Have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of ranolazine.
3. Documented hypersensitivity to any component of ranolazine (Ranexa®) pills.
4. Need for medications that are:

   1. strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors (e.g. ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, saquinavir),
   2. moderate CYP3A inhibitors (e.g. diltiazem, verapamil, erythromycin, fluconazole, grapefruit juice or grapefruit-containing products),
   3. CYP3A inducers (e.g. rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, St. John's wort),
   4. CYP3A substrates with a narrow therapeutic range (e.g. cyclosporine, tacrolimus, sirolimus),
   5. P-gp inhibitors or substrates (e.g. cyclosporine, digoxin),
   6. polypeptide 6 (CYP2D6) substrates (e.g. tricyclic antidepressants and antipsychotics),or
   7. simvastatin at doses > 20 mg/day.
5. Have corrected QT interval (QTc)> 450 msec (male) or > 470 msec (female) on 12-lead electrocardiogram.
6. Poorly controlled diabetes, hemoglobin A1c (Hgb A1C) >9 or random blood glucose >250mg/dL.
7. Active or symptomatic viral hepatitis or chronic liver disease.
8. Clinically significant heart disease as evidenced by:

   1. myocardial infarction, or
   2. arterial thrombotic events in the past 6 months,
   3. severe or unstable angina, or
   4. New York Heart Association Class III-IV heart disease or
   5. cardiac ejection fraction measurement of <50%.
9. Active infection requiring antibiotics.
10. Major surgery or radiation treatment within 3 months.
11. Cytotoxic chemotherapy within 4 weeks.
12. Immunotherapy within 6 months.
13. Any prior therapy with Radium-223, Samarium, or Strontium.
14. Arm 1 patients may not have received any prior luteinizing-hormone-releasing hormone (LHRH) agonists/antagonists, anti-androgens, or chemotherapy for their prostate cancer. 5-alpha reductase inhibitors (finasteride, dutasteride) may be allowed.
15. Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2016-10-08 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Lam, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Localized Prostate Cancer) | Arm II (Metastatic Prostate Cancer)
Started | 4 | 7
Completed | 4 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Localized Prostate Cancer) | Arm II (Metastatic Prostate Cancer) | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 7 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Increase in SUV Uptake
Description: Number of participants who had increased SUV uptake, as defined by any of the following:
  1. SUVmax increase of 30% with a 2 unit absolute change.
  2. SUVmean increase of 30% with a 0.75 unit absolute change.
  3. SUVmean increase of 20% with a 1 unit absolute change.
Time Frame: Within 1 week after completion of ranolazine treatment
Population: This study was closed to accrual early. Due to small numbers, no statistical or firm conclusions can be made on the basis of such small numbers.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Localized Prostate Cancer) | Arm II (Metastatic Prostate Cancer)
Number analyzed (Participants) | 4 | 7
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse effects to the ranolazine for the duration of the study which lasted from screening to completion of prostatectomy (Arm I; about 8 weeks) or completion of PET/CT (Arm II; about 4 weeks).
Arm/Group | Arm I (Localized Prostate Cancer) | Arm II (Metastatic Prostate Cancer)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No